CLINICAL TRIAL: NCT03954808
Title: The Effect of Motor Imagery Training on Muscle Activity, Motor Imagery and Functional Movement Skills in Individuals Unilateral Cerebral Palsy
Brief Title: Motor Imagery Training in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Demet Karabulut, PhD Student, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbantIBU-FTR-DK-1
Record Dates: First submitted 2019-05-16; First posted 2019-05-17 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Palsy
Keywords: Unilateral Cerebral Palsy, Motor imagery,
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery training group (Experimental): Children with Cerebral Palsy. Motor imagery training group will receive a traditional physiotherapy and motor imagery training within a specific program, two days a week for a total of 8 weeks (30 minutes traditional physiotherapy session+15 minutes MI training). The motor imagery training will be designed for the individual basis with standard protocols. All sessions will be performed in the clinic.
  Interventions: Other: Motor Imagery Training
- Cerebral Palsy control group (Active Comparator): Children with Cerebral Palsy. Traditional physiotherapy control group individuals will be given a traditional physiotherapy two days per week for a total of 8 weeks (traditional physiotherapy session will last 45 minutes).
  Interventions: Other: Traditional physiotherapy
- Typically developing control group (No Intervention): Age matched healthy individuals, with no treatment.

INTERVENTIONS:
Other: Motor Imagery Training — Motor imagery training will be designed for the individual basis with standard protocols
  Arms: Motor imagery training group
Other: Traditional physiotherapy — Traditional physiotherapy within a specific program
  Arms: Cerebral Palsy control group

SUMMARY:
Motor imagery (MI) is a promising method to improve more cognitive aspects of motor behaviour, and may, thus, be effective for facilitating motor planning in children with Cerebral Palsy (CP). MI training facilitates the neural plasticity by enhancing the neuronal cortical pathways in brain. In children with CP, motor planning and MI capacity were found to be affected by studies. In the literature, there are studies about the evaluation of MI in Unilateral CP but there is insufficient number of studies included in MI in the rehabilitation program.

The aim of the study was to investigate the effect of motor imagery training for gait and lower extremity muscle activity (with EMG), functional capacity, quality of life, and time performance variables in Children with Unilateral CP.

The eligible participants will be allocated three groups, including motor imagery training group, traditional physiotherapy control group, and healthy control group. All the assessments will be performed before and after the training in the 8-week motor imagery training group and 6 weeks after the end of training. The participants in the control group will be evaluated with a 8-week interval and 6 weeks after the end of physiotherapy training. The healthy participants will be assessed only once. The motor imagery training will be designed for the individual basis with standard protocols. It will be applied two times a week for 8 weeks. All sessions will be performed in the clinic.

DETAILED DESCRIPTION:
Unilateral CP and age matched healthy individuals will be participate the study between the ages of 7 and 18 years. Children's gross motor skills classified with GMFCS.

The control group individuals will be given a traditional physiotherapy two days per week for a total of 8 weeks (traditional physiotherapy session will last 45 minutes). Motor imagery training group will receive a traditional physiotherapy and motor imagery training within a specific program, two days a week for a total of 8 weeks (30 minutes traditional physiotherapy session+15 minutes MI training) .

Within the scope of MI training, individual training program will be determined by taking into consideration the needs of the individuals and the expectations for gait. The basic case of PETTLEP (Physical, Environment, Task, Timing, Learning, Emotion, Perspective) will be followed. MI training will be given individually with the same physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cerebral Palsy voluntary participation
* Age between 7-18 years, Children with Unilateral Cerebral Palsy
* With suitable cognitive state for training
* To attend a formal school
* GMFCS Level I-II
* IQ>70 Children with Unilateral Cerebral Palsy (from children's file)
* Mini-Mental State Exam For Children score above 24

Exclusion Criteria:

* Severe cognitive impairment and not able to follow task instructions
* IQ<70 Children with Unilateral Cerebral Palsy (from children's file)
* Who received motor imagery training last 6 months
* Severe Vision and hearing problems
* Botox or surgeries in the last 6 months

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Movement Imagery Questionnaire-Children(MIQ-C) | Change from Baseline at 8 weeks and 14 weeks
  Visual and Kinesthetic motor imagery ability will be evaluated with MIQ-C. Includes 12 items in total. The individual is asked to visualize four different movements from three different imagery perspectives. The clearness of the imagination is scored using a Likert-type scale between 1 (very difficult to feel) -7 (very easy to feel)
Mental Chronometry for Timed Up and Go Test | Change from Baseline at 8 weeks and 14 weeks
  Motor imagery capacity will be evaluated by mental chronometry. This paradigm compares the duration between the actual movement and the imagined movement similar task duration. In this paradigm, participants are asked to do the Timed Up and Go test (TUG) and then they are asked to imaging the TUG. The timing of the imaging and actual movement will be determined by the stopwatch. Then compare the duration of actual and imagined movements. The temporal accuracy between actual and imagined movement will be calculated in terms of the delta time.

SECONDARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | At Baseline
  Assessing severity of the disability and motor function. Gross motor functions of children with CP are classified in five levels with GMFCS. This is a classification system based on the child's self-initiated movements with emphasis on sitting, displacement and mobility.
Modified Tardieu Scale (MTS) | Change from Baseline at 8 weeks and 14 weeks
  Assessing muscle tone of individuals. It evaluates reaction of the muscle to passive movement of limb both slow and fast speeds. This scale evaluated the speed-dependent nature of spasticity. Quality of muscle reaction (X) and the angle of muscle reaction (Y) are determined by the modified tardieu scale. If quality of muscle reaction score was 2 or higher, the joint angle in which the muscle responds with difficulty will be measured goniometer. The Modified Tardieu Scale scores range from 0 to 5. Scoring: 0= no resistance to passive movement. 1= slight resistance throughout the course of the passive movement. 2= there's a clear catching at a precise angle, which makes passive movement difficult, followed by a release. 3= fatigable clonus (Less than 10 seconds). 4= infatigable clonus (More than 10 seconds). 5= the joint cannot be moved.
Conner's Parent Rating Scale-Revised Short form (CPRS-RS) | At Baseline
  Assessing whether individuals' levels of attention differ from between groups. The questionnaire consisted of 27 items and three sub-dimensions (Oppositionality, Hyperactivity, Cognitive Problems-Inattention). Response formats are in the form of a four-point Likert type scale. Answer options and scoring are as follows: 0 points are never correct, 3 points are very accurate, with total scores ranging from 0 to 81. Cognitive Problems-Inattention subscale has the minimum score is 0 and the maximum score is 18. Higher scores are reflective of worse situations of attention.
Mini-Mental State Exam For Children (Mmc) | At Baseline
  Mini-Mental State Exam For Children (Mmc) consists of 15 questions designed to assess the cognitive functions of the individual. Includes recording, recall, attention and calculation, temporal orientation, spatial orientation, and language measurement. It takes about 15 minutes to perform.
Surface electromyography (sEMG) | Change from Baseline at 8 weeks and 14 weeks
  Surface electromyography is a non-invasive method that involves taking, recording and interpreting the electric activity of muscle groups. Delsys Trigno Wireless System superficial EMG (sEMG) device will be used for evaluation of muscle activation. Measurements will be made in accordance with the criteria of SENIAM (surface EMG for non-invasive assessment of muscle) and the literature. Activation of lower extremity muscles through silver-silver chloride (Ag-AgCl) disposable adhesive electrodes will be evaluated.
Pediatric Evaluation of Disability Inventory (PEDI) | Change from Baseline at 8 weeks and 14 weeks
  Assessing disability and activity and participation. 0: can not do, 1: can do in the form of scoring is done. At the end of the evaluation, the points of the related section are collected.
Pediatric Outcomes Date Collection (PODCI) (Questionnaire) | Change from Baseline at 8 weeks and 14 weeks
  Assessing health-related quality of life, activity and participation. It consists of five basic sub-groups; upper extremity functions, physical function and sport, transfer and base mobility, pain, happiness / satisfaction.
Timed Up and Go Test | Change from Baseline at 8 weeks and 14 weeks
  The Timed Up and Go test (TUG) is a simple test used to assess functional mobility, dynamic balance, walking speed and postural stability. The individual is asked to rise from chair, walk three meters safe and normal speed, turn around, walk back to the chair and sit down. The time is calculated in seconds from the start of the instruction to ends when the patient is seated.
10-Meter Walk Test | Change from Baseline at 8 weeks and 14 weeks
  The individual is asked to walk the distance of 10 meter three times with the maximum speed that he or she wants can walk and the average time is recorded.
Five Times Sit to Stand Test | Change from Baseline at 8 weeks and 14 weeks
  This test is associated with lower extremity muscle strength and balance. During the test, the individual is asked to stand up and sit for five times without holding up from the chair and the elapsed time is recorded.
Mental Chronometry for 10-Meter Walk Test | Change from Baseline at 8 weeks and 14 weeks
  Motor imagery capacity is evaluated by mental chronometry. This paradigm compares the duration between the actual movement and the imagined movement similar task duration. In this paradigm, participants are asked to do the 10-Meter Walk Test and then they are asked to imaging the this test. The timing of the imaging and actual movement will be determined by the stopwatch. Then compare the duration of actual and imagined movements. The temporal accuracy between actual and imagined movement will be calculated in terms of the delta time.
Mental Chronometry for Five Times Sit to Stand Test | Change from Baseline at 8 weeks and 14 weeks
  Motor imagery capacity is evaluated by mental chronometry. This paradigm compares the duration between the actual movement and the imagined movement similar task duration. In this paradigm, participants are asked to do the Five Times Sit to Stand Test and then they are asked to imaging the this test. The timing of the imaging and actual movement will be determined by the stopwatch. Then compare the duration of actual and imagined movements. The temporal accuracy between actual and imagined movement will be calculated in terms of the delta time.
Laterality Task | Change from Baseline at 8 weeks and 14 weeks
  This task evaluates the left-right discrimination and implicit imagery. Two aspects will be evaluated in the task of recognition of the foot's laterality. First, the precision (percentage of right answers) of the discrimination of the laterality which is the capacity to recognize whether a part of the body belongs to the right or left and second the response time of the participants use in the discrimination task. NOI group designed and developed application about this will be used.
Functional muscle strength | Change from Baseline at 8 weeks and 14 weeks
  The 30s Repetition Maximum test will be used to assess functional muscle strength of the lower extremities. The three closed kinetic chain exercises of lateral step-up test, sit to stand test, and attain stand through half knee test will be used.
Motor imagery entertainment scale | Change from Baseline at 4 weeks and 8 weeks
  The entertainment level of motor imagery sessions and imagery training for individuals will be evaluated with a 0-10 point numerical rating scale (entertainment scale). There are numbers from 0 to 10 on the horizontal line of 10 cm. 0 "Not fun" on the line in the scale; 10 represents "a lot of fun". Entertainment rating will be recorded numerically from 0 to 10.
Motor imagery clarity scale | Change from Baseline at 4 weeks and 8 weeks
  The clarity level of motor imagery sessions and imagery training for individuals will be evaluated with a 0-10 point numerical rating scale (clarity scale). There are numbers from 0 to 10 on the horizontal line of 10 cm.
  On the horizontal 10 cm horizontal line, 0 means that the visualization never occurs, and 10 indicates that it is very clear. Clarity rating will be recorded numerically from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem T Yümin, Study Director — Abant Izzet Baysal University
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steenbergen B, Craje C, Nilsen DM, Gordon AM. Motor imagery training in hemiplegic cerebral palsy: a potentially useful therapeutic tool for rehabilitation. Dev Med Child Neurol. 2009 Sep;51(9):690-6. doi: 10.1111/j.1469-8749.2009.03371.x. PMID 19709140
- [Background] Steenbergen B, Jongbloed-Pereboom M, Spruijt S, Gordon AM. Impaired motor planning and motor imagery in children with unilateral spastic cerebral palsy: challenges for the future of pediatric rehabilitation. Dev Med Child Neurol. 2013 Nov;55 Suppl 4:43-6. doi: 10.1111/dmcn.12306. PMID 24237279
- [Background] Lust JM, Wilson PH, Steenbergen B. Motor imagery difficulties in children with Cerebral Palsy: A specific or general deficit? Res Dev Disabil. 2016 Oct;57:102-11. doi: 10.1016/j.ridd.2016.06.010. Epub 2016 Jul 9. PMID 27399206

DOCUMENTS (2):
  • Study Protocol (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03954808/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT03954808/SAP_001.pdf